CLINICAL TRIAL: NCT00927316
Title: Induced Asymptomatic E. Coli 83972 Bacteriuria in Patients With Recurrent Urinary Tract Infections and Bladder Dysfunction- is There a Protective Effect Against Recurrent Symptomatic Infections? A Blinded Placebo Controlled Cross-over Study.
Brief Title: E. Coli 83972 Induced Asymptomatic Bacteriuria (ABU) in Patients With Recurrent Urinary Tract Infections (UTI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Coloplast A/S (Industry); Riksförbundet för Trafik, Olycksfall och Polioskadade (RTP), Sundbyberg, Sweden (Unknown); Swedish Institute for Infectious Disease Control (Other); Lund University Hospital (Other)
Responsible Party: Fredrik Sundén, MD, Dept. of Urology, University Hospital, Lund, Sweden
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: RTP-A2003
Record Dates: First submitted 2009-06-22; First posted 2009-06-24 (Estimated); Last update posted 2009-11-10 (Estimated); Status verified 2009-11

CONDITIONS: Urinary Tract Infection
Keywords: Report of Urinary Tract Infection episode
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active arm (Active Comparator): E. coli 83972 bacteriuria
  Interventions: Biological: E. coli 83972
- Placebo arm (Placebo Comparator): Monitoring
  Interventions: Biological: E. coli 83972

INTERVENTIONS:
Biological: E. coli 83972 — Active arm: Intravesical inoculation (by urethral catheterization) on three subsequent days with 30 ml E. coli 83972 (100 000 cfu/ml).
  Placebo arm: Identical procedure but with saline, 30 ml.

SUMMARY:
This study tests the following hypothesis: Does induced asymptomatic bacteriuria (E. coli 83972) protect against symptomatic urinary tract infections in individuals with bladder emptying dysfunctions and prone to recurrent infection episodes? The study is performed using a double-blind randomized study protocol with a cross-over, with re-inoculations being patient-blinded (phase 1). After patients have fulfilled the cross-over, those who have had bacteriuria or placebo-periods < 12 months will be subjected to additional patient blinded inoculations (phase 2). During the entire study (phase 1+2) the study-team and the patients are unaware of urine culture results.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent UTI
* Bladder emptying dysfunction
* Optimal conservative treatment incl. clean intermittent catheterization
* Capable of "self reporting of UTI episodes"

Exclusion Criteria:

* Malignant disease
* Immunosuppression
* Recurrent pyelonephritis
* Abnormalities within upper urinary tract, including renal stones and poor kidney function

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2003-03; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Time to UTI | 12 months
Number of UTI | During 12 months placebo or active treatment

CONTACTS AND LOCATIONS:
Overall Officials: Fredrik Sundén, MD, Principal Investigator — Dept. of Urology, University Hospital, 221 85 Lund; Björn Wullt, MD, PhD, Study Chair — Dept. of Urology, Lund University Hospital, 221 85 Lund
Locations (1):
- Department of Urology, Lund University, Lund, Sweden